CLINICAL TRIAL: NCT05295953
Title: Accelerated Transcranial Magnetic Stimulation (TMS) for Smoking Cessation in People Living With HIV/AIDS (PLWHA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 70889; 5P30CA177558-10 (NIH)
Record Dates: First submitted 2022-02-10; First posted 2022-03-25 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Hiv; Tobacco Smoking
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: Active group and sham group
Who Masked: Participant, Care Provider
Masking Description: Participant will not know whether they receive active or sham TMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- TBS (Theta burst stimulation) (Active Comparator): Four sessions of TBS in one day
  Interventions: Device: TBS
- Sham TMS (Placebo Comparator): Four sessions of sham TMS
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: TBS — Four sessions of TBS at 120 % resting motor threshold, delivered using MagVenture B65 A/P coil, each lasting 10 minutes and separated by 50 minutes intervals. Targeting will be done using neuronavigation and processed resting state brain scan.
  Arms: TBS (Theta burst stimulation)
Device: Sham TMS — Four sessions of sham TMS delivered using MagVenture B65 A/P coil.
  Arms: Sham TMS

SUMMARY:
To demonstrate whether four sessions of TBS improves attentional bias and craving in PLWHA smokers compared to four sessions of sham stimulation. We hypothesize 4 sessions of TBS to the left DLPFC will significantly improve attentional bias and craving for smoking cues compared to neutral cues in a population of subjects who are smokers with HIV/AIDS compared to sham stimulation.

DETAILED DESCRIPTION:
The proposed pilot study seeks to explore modulation of attentional bias and tobacco craving in PLWHA with one session of adequately dosed theta burst stimulation (TBS). Results of this trial will spur clinical research to further investigate the use of TBS as an adjunctive smoking cessation aid for PLWHA and could have broad implications for smoking cessation programs. Data obtained from this pilot study will also facilitate resubmission of a grant application examining adjunctive theta burst stimulation (TBS) combined with varenicline for smoking cessation in PLWHA. People living with HIV/AIDS (PLWHA) smoke at nearly three times the rate of the general population. These extraordinary smoking rates are associated with greater AIDS-related morbidity, non-AIDS related morbidity including non-AIDS-defining cancer, cardiovascular disease, pulmonary disease, and mortality. Smoking significantly impacts the progression and outcome of HIV disease and has been identified as the leading contributor to premature mortality in PLWHA. One study estimated PLWHA lose more years from smoking than from HIV infection. In our view, shared by others in the field, the single greatest health behavior change that could improve mortality is to assist smokers living with HIV/AIDS to quit smoking.

ELIGIBILITY:
Inclusion Criteria: Potential participants will be

* Patients enrolled in the Bluegrass Clinic
* 18-60 years of age
* Male or female gender
* Able to read, understand and communicate in English
* Willing to adhere to the general rules of the Bluegrass Clinic/SMARTClinic/Beyond Birth Clinic
* Willing and able to abstain from drug use other than Suboxone
* Exhaled breath on day of study carbon monoxide (CO) < 5 ppm
* Stabilized on maintenance buprenorphine if having comorbid opioid use disorder.

Exclusion Criteria:

* Positive pregnancy test for females, traumatic brain injury, history of seizure disorder, history of or current diagnosis of schizophrenia, intracranial metal shrapnel.
* Previous adverse effect with TMS.
* Sub-threshold consistency while performing behavioral tasks.
* Failure to show baseline attentional bias to smoking versus neutral cues.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - 245 Fountain Court, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky

REFERENCES:
- [Derived] Rakesh G, Alcorn JL 3rd, Khanal R, Himelhoch SS, Rush CR. Comparing cigarette-cue attentional bias between people with HIV/AIDS and people with opioid use disorder who smoke. Health Psychol Behav Med. 2023 Sep 7;11(1):2255028. doi: 10.1080/21642850.2023.2255028. eCollection 2023. PMID 37693107

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (10.6) | 40.7 (1.4) | 45.25 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Gaze Fixation on Smoking Cues
Description: Measured using an eye tracker which quantifies this in milliseconds, higher score means worse outcome
Time Frame: On Day 1 of the study
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
Number analyzed (Participants) | 2 | 1
milliseconds | 320.19 (234.83) | 152.60 (NA) — ONLY ONE PARTICIPANT DATA ANALYZED

2. Primary Outcome: Gaze Fixation on Smoking Cues
Description: Measured using an eye tracker which quantifies this in milliseconds, higher score means worse outcome
Time Frame: On Day 1 of the study after intervention
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
Number analyzed (Participants) | 2 | 1
milliseconds | 221.75 (94.24) | 120.50 (NA) — Only one participant's data analyzed

3. Primary Outcome: Craving for Cigarettes
Description: Measured using tobacco craving questionnaire (TCQ), this questionnaire has 12 items. Max score is 84, min score is 0. Higher score means that craving is higher.
Time Frame: On day one of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
Number analyzed (Participants) | 2 | 1
units on a scale | 58 (5.66) | 50 (NA) — Only one participant's data analyzed

4. Primary Outcome: Craving for Cigarettes
Description: as for outcome 3
Time Frame: Immediately after intervention (sessions of TBS or sham TMS) on day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
Number analyzed (Participants) | 2 | 1
units on a scale | 51 (1.41) | 28 (NA) — Only one participant's data analyzed

5. Secondary Outcome: Number of Participants Showing Functional Connectivity Changes
Description: Changes in functional connectivity on a functional MRI brain scan.
Time Frame: on Day 1 of study
Measure: Count of Participants; unit: Participants
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
Number analyzed (Participants) | 2 | 1
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TBS (Theta Burst Stimulation) | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT05295953/Prot_SAP_001.pdf
  • Informed Consent Form (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT05295953/ICF_000.pdf